CLINICAL TRIAL: NCT03717519
Title: Elevated Platelet Count as Prognostic Factor in Colorectal Cancer With Synchronous Liver Metastases: a Retrospective Single-center Cohort Study
Brief Title: Elevated Platelet Count as Prognostic Factor in Colorectal Cancer With Synchronous Liver Metastases
Acronym: PLTCRC
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Corrado Pedrazzani, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: CHIR CR
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Stage IV Colon Cancer
Keywords: platelets; thrombocytosis; prognosis
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Thrombocytosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- s-CRLM: Patients with synchronous colorectal liver metastases who underwent surgical resection
  Interventions: Diagnostic Test: Measurement of platelet count at diagnosis

INTERVENTIONS:
Diagnostic Test: Measurement of platelet count at diagnosis — Blood samples were drawn by expert phlebotomists in vacuum blood tubes containing K2-EDTA (Terumo Europe NV, Leuven, Belgium). The complete blood cell count (CBC) was performed using Advia 2120 (Siemens Healthcare Diagnostics, Tarrytown NY, USA). The local reference range for platelets was 150-400 x 109/L. The same analyser was used throughout the study period, and the quality and reproducibility of test results was validated by data of both internal quality control and external quality assessment

SUMMARY:
Colorectal cancer (CRC) is the third most common malignancy worldwide and is often metastatic at diagnosis. Despite progresses in surgical techniques and the introduction of novel chemotherapy regimens, many patients still suffer from a poor prognosis. It is therefore of utmost importance to identify prognostic markers that may improve selection of patients.

In recent years several studies demonstrated that preoperative blood tests as platelet count or neuthophil-to-lymphocyte ratio could be prognostic factors in CRC as well as other malignancies. The aim of this study was to evaluate the role of preoperative platelet count (PC) in patients with synchronous colorectal liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer with synchronous liver metastases
* Possibility to retrieve pre-operative platelet count
* Age of 18 years or older
* Availabilty of clinical-pathological data
* Minimum follow up of 12 months

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgery for colorectal cancer with synchronous liver metastases in the study period, and who fulfilled the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
  correlation between high PC and overall survival

SECONDARY OUTCOMES:
Clinic-pathological variables | 30 days
  correlation between high PC and clinic-pathological variables

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Pedrazzani, MD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona
Locations (1):
- Chirurgia Generale ed Epatobiliare, Policlinico GB Rossi, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pedrazzani C, Mantovani G, Fernandes E, Bagante F, Luca Salvagno G, Surci N, Campagnaro T, Ruzzenente A, Danese E, Lippi G, Guglielmi A. Assessment of neutrophil-to-lymphocyte ratio, platelet-to-lymphocyte ratio and platelet count as predictors of long-term outcome after R0 resection for colorectal cancer. Sci Rep. 2017 May 4;7(1):1494. doi: 10.1038/s41598-017-01652-0. PMID 28473700
- [Background] Wan S, Lai Y, Myers RE, Li B, Hyslop T, London J, Chatterjee D, Palazzo JP, Burkart AL, Zhang K, Xing J, Yang H. Preoperative platelet count associates with survival and distant metastasis in surgically resected colorectal cancer patients. J Gastrointest Cancer. 2013 Sep;44(3):293-304. doi: 10.1007/s12029-013-9491-9. PMID 23549858
- [Background] Baranyai Z, Krzystanek M, Josa V, Dede K, Agoston E, Szasz AM, Sinko D, Szarvas V, Salamon F, Eklund AC, Szallasi Z, Jakab F. The comparison of thrombocytosis and platelet-lymphocyte ratio as potential prognostic markers in colorectal cancer. Thromb Haemost. 2014 Mar 3;111(3):483-90. doi: 10.1160/TH13-08-0632. Epub 2013 Nov 28. PMID 24285160